CLINICAL TRIAL: NCT03207126
Title: Pilot Study: Can Ultrasound Guided Biopsy be Used as an Alternative to Hysteroscopy in the Detection of Endometrial Cancer?
Brief Title: Pilot Study: Can Ultrasound Guided Biopsy be Used as an Alternative to Hysteroscopy?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16HH3687 USS guided biopsy EC
Record Dates: First submitted 2017-06-30; First posted 2017-07-02 (Actual); Results first posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-10

CONDITIONS: Endometrial Cancer; Endometrial Neoplasms; Endometrial Hyperplasia; Endometrial Polyp
Keywords: Ultrasound; Biopsy; Endometrial cancer
MeSH Terms: conditions — Endometrial Neoplasms; Endometrial Hyperplasia

STUDY DESIGN:
Intervention Model Description: Women offered and received ultrasound guided biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Women needing endometrial biopsy (Other): All women who would be offered hysteroscopy guided biopsy as standard of care will be offered ultrasound guided biopsy first.
  Interventions: Diagnostic Test: Ultrasound guided biopsy

INTERVENTIONS:
Diagnostic Test: Ultrasound guided biopsy — For women needed a hysteroscopy guided biopsy as part of routine standard of care, women will now receive an ultrasound guided biopsy first

SUMMARY:
Aim: Assess accuracy of histological diagnosis using ultrasound guided biopsy for women with suspected endometrial cancer (as an alternative to hysteroscopy guided biopsy).

All women presenting to clinic with suspected endometrial cancer will have an internal ultrasound. If the endometrial lining is thickened an endometrial biopsy will be performed. This can sometimes be done in an outpatient clinic, or sometimes a hysteroscopy and biopsy is needed (on a different day). Hysteroscopy guided biopsy has the advantage of enabling the clinician to perform directed biopsies under vision.

Ultrasound guided biopsy is a ubiquitous procedure when used elsewhere in the body however it is not routinely used in this context. It does have the advantage of being easily performed on the same day as the first consultation. In this pilot study the diagnostic ability and tolerability of ultrasound guided biopsy of women with suspected cancer will be assessed as an alternative to hysteroscopy guided biopsy.

DETAILED DESCRIPTION:
Aims: Assess accuracy of histological diagnosis using ultrasound guided biopsy for women with suspected endometrial cancer (as an alternative to hysteroscopy guided biopsy).

Background:

Endometrial cancer is a tumour originating in the endometrium (womb lining); it is the most common gynaecological cancer in the UK. Although routine management for these women does vary, in general a screening test is performed, typically a pelvic (internal) ultrasound to assess the endometrium (womb lining). In cases where the endometrial thickness is above the threshold for investigation - an endometrial biopsy (sampling cells from the womb lining) is indicated. The biopsy can be taken blindly or under scan or hysteroscopic guidance. Hysteroscopy, the insertion of a small camera into the womb to visualise the womb lining allows direct visualization of the cavity. This usually occurs at a separate consultation in an outpatient setting or under general anaesthesia.

In theory an ultrasound-guided biopsy using a very fine Bettocchi forceps could be used instead of hysteroscopy- guided biopsies of the endometrium. The technique of ultrasound-guided biopsy is ubiquitous when used elsewhere in the body. It is frequently used to provide histological diagnosis of pelvic masses, (presumed ovarian origin), both abdominally (scanning of the tummy) and transvaginally (internally). Potentially ultrasound guided biopsies could be used as a cheaper, faster and less painful alternative to a hysteroscopy directed biopsies. This pilot study will be the first to assess the diagnostic ability of ultrasound guided biopsy in the assessment of women with suspected endometrial cancer.

The study:

All women will receive a pelvic (internal) ultrasound as per routine care. If the endometrium (womb lining) is thickened >4mm on ultrasound they will require an endometrial biopsy. Usually this will be a pipelle. In cases where the pipelle biopsy cannot be performed in clinic due to poor tolerance, insufficient material or focal lesions a hysteroscopy guided biopsy will be required (local or GA).

In this case, the patients will be offered an ultrasound (USS) guided biopsy in the first instance, this will be performed at the same time in clinic. The biopsy will be taken under scan guidance using a very fine forceps such as Bettochi forceps. These forceps are used routinely during hysteroscopy so whilst the instruments are common the application is novel. The biopsy results of this will be sent for standard histology. If the results are inadequate patients will be sent for standard hysteroscopy and biopsy. Patients will also be asked to assess tolerability of the procedure using a visual analogue score.

ELIGIBILITY:
Inclusion Criteria:

All women presenting to rapid access gynaecology clinic with postmenopausal bleeding or intermenstrual bleeding or referred with a confirmed diagnosis of endometrial cancer.

Exclusion criteria:

Anyone lacking capacity. <18years old. Pregnant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Study is looking at endometrial cancer
Enrollment: 10 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana Marcus, MB BS, Principal Investigator — Imperial College London
Locations (1):
- Queen Charlotte and Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Will share results if published only.

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: samples
Period: Overall Study
Arm/Group | Women Needing Endometrial Biopsy
Started | 10; 10 samples
Completed | 10; 10 samples
Not Completed | 0; 0 samples

BASELINE CHARACTERISTICS:
Arm/Group | Women Needing Endometrial Biopsy
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 4
Age, Continuous [Median (Full Range); unit: years] | 61 [45 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 10
Pain score [Median (Inter-Quartile Range); unit: units on a scale] — The pain score range was 0 to 10 where 0 means low pain and 10 worst pain ever had.
  units on a scale | 7.5 [6 to 10]
Number of participants providing a tissue sample [Count of Participants; unit: Participants] — The sample was taken using ultrasound and tested thereafter using histology.
  Participants | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Whose Sample Was Successfully Analysed by Histological Diagnosis
Description: All samples taken using ultrasound guided biopsy were analysed by histology lab. If they had sufficient tissue to give a diagnosis (benign, pre-malignant or malignant) this was deemed successful. It is deemed successful if there was sufficient tissue to give a histological analysis. So overall there will be a percentage success rate (number of tissue samples sufficient/number of tissue samples taken). Each patient would have had one sample.
Time Frame: 1.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Women Needing Endometrial Biopsy
Number analyzed (Participants) | 10
Participants | 9

2. Secondary Outcome: Patient Satisfaction of Ultrasound Guided Biopsy by Questionnaire
Description: Visual analogue score will be given to patients post procedure to assess tolerability of the procedure. The full score scale ranges from 0 to 10 that means from no pain (0) to worst pain they ever had (10).
Time Frame: 1.5 years
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Women Needing Endometrial Biopsy
Number analyzed (Participants) | 10
score on a scale | 7.5 [4 to 10]

ADVERSE EVENTS:
Time Frame: 1.5 years
Description: Please see below.
Arm/Group | Women Needing Endometrial Biopsy
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-07-14): https://cdn.clinicaltrials.gov/large-docs/26/NCT03207126/Prot_SAP_000.pdf